CLINICAL TRIAL: NCT05803083
Title: The Effect of Oral Hyaluronic Acid on the Skin-A Randomized-Blind, Placebo-Controlled Study-
Brief Title: The Effect of Oral Hyaluronic Acid on the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloomage Biotechnology Corp., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-2023-BMB01
Record Dates: First submitted 2023-03-02; First posted 2023-04-07 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-03

CONDITIONS: Healthy Japanese Subjects
Keywords: Hyaluronic Acid; Skin
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic Acid 150 mg (Active Comparator): Take 150 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: Hyaluronic acid 75 mg/capsule
- Hyaluronic Acid 100 mg (Active Comparator): Take 100 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: Hyaluronic acid 50 mg/capsule
- Placebo (Placebo Comparator): Take 0 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hyaluronic acid 75 mg/capsule — Take 2 capsules per day at any time.
  Arms: Hyaluronic Acid 150 mg
Dietary Supplement: Hyaluronic acid 50 mg/capsule — Take 2 capsules per day at any time.
  Arms: Hyaluronic Acid 100 mg
Dietary Supplement: Placebo — Take 2 capsules per day at any time.
  Arms: Placebo

SUMMARY:
This clinical trial aims to clarify the effect of hyaluronic acid on skin conditions.

DETAILED DESCRIPTION:
In this study, investigators will evaluate the skin condition before and after the intervention. The groups to be compared are two different doses of hyaluronic and a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese women between 30 and 60 years of age at the time of obtaining consent to participate in the study.
2. Healthy individuals with no chronic physical diseases, including skin diseases.
3. Person with sagging, dry, or flaky skin.
4. Person who have been fully informed of the purpose and content of the study, have the capacity to consent, understand it well, and voluntarily volunteer to participate in the study, and are able to consent to participation in the study in writing.
5. Person who be able to come to the study site on the designated examination date and undergo the examination.
6. Person who are deemed suitable by the investigator to participate in the study.

Exclusion Criteria:

1. Those who currently suffer from some disease and are receiving drug treatment.
2. Patients with skin disease symptoms such as atopic dermatitis.
3. Patients who have scars or inflammation on the evaluation site.
4. Patients who have taken or applied drugs in the past month for the purpose of treatment of the disease (excluding those who have taken drugs for headache, menstrual cramps, common cold, etc.).
5. Patients with a history or current history of serious disorders of the liver, kidney, heart, lungs, blood, etc.
6. Patients with comorbidities and serious history of gastrointestinal disorders.
7. Patients with severe anemia.
8. BMI of 30.0 kg/m2 or more.
9. Person who are allergic to any ingredient in the test food or who are at risk of developing serious allergic reactions to any other food or drug.
10. person is currently, or within the past 3 months has been, or will be during the study period, a habitual consumer of functional foods, health foods, or supplements containing active ingredients similar to those in the test food.
11. Currently, and within the past 3 months, those who have or will take functional foods, health foods, or supplements that claim to improve skin on a regular basis during the study period (consumption for the purpose of maintaining good health is acceptable).
12. Currently, or within the past 3 months, those who have a habit of continuously taking or applying drugs that are claimed to improve the skin.
13. Pregnant, lactating, or of child-bearing potential.
14. Patients whose daily alcohol consumption exceeds an average of 60g/day of pure alcohol equivalent.
15. Patient with mental disorders.
16. Persons with a smoking habit.
17. Those who may change their lifestyle during the examination period (e.g., work at night, travel for long periods of time, etc.).
18. Patient who may develop seasonal allergic symptoms such as hay fever and may use medicines during the study period.
19. Persons who will be extremely neglectful of their skin care.
20. Those who intentionally cannot refrain from being exposed to direct sunlight, such as sunburn, during the examination period.
21. Person with a history of cosmetic procedures or treatments on the evaluation site within the past 6 months.
22. Person with currently participating in another human clinical trial, or who have not yet completed 3 months of participation in another human clinical trial.
23. Person who are judged by the investigator to be inappropriate for this study.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin viscoelasticity | Week0, 2, 4, 8 and week 4 after the end of intake
  In skin viscoelasticity measurement using Cutometer MPA580®, skin displacement is measured by applying negative pressure to the skin through the opening of the probe and releasing the negative pressure. The higher the value, the greater the viscoelasticity.
  Measurement part：Measure the center of the left face, connecting the bottom of the earlobe and the edge of the lip.
  Accepted value：Measure the same place 5 times, and use the average of 3 measurements with the highest and lowest value data removed based on the R2 value.
  Analysis target value：R0, R2, R5, R7

SECONDARY OUTCOMES:
Change from baseline skin moisture content | Week0, 2, 4, 8 and week 4 after the end of intake
  Skin moisture content is evaluated by using a Corneometer CM825®t
Change from baseline trans-epidermal water transpiration | Week0, 2, 4, 8 and week 4 after the end of intake
  Trans-epidermal water transpiration is evaluated by using Tewameter TM300®
Change from baseline VISIA image | week 0, 2, 4, 8 and week 4 after the end of intake
  Analyze the following items are measured and simply by putting face into VISIA Evolution.
  Measurement points：Photograph the left face Analysis target value：Blemishes, Wrinkles, Texture. Pores, Ultraviolet Blemishes, Brown Blemishes, Red Areas, Porphyrin.Higher numbers for these items indicate more advanced aging.
  Gloss is measured by VISIA-CR.
Change from baseline face visual evaluation | Week0, 2, 4, 8 and week 4 after the end of intake
  Face visual evaluation is measured by the dermatologist. Evaluation items：Cutaneous carpus, cutaneous groove, comprehensive evaluation Evaluation site：Evaluation centered on the left face, connecting the lower earlobe and the edge of the lip Evaluation method：Perform visual judgment using DermLite DL100 (J Hewitt Co., Ltd.) and microscope (KH-1300/HXG-2016Z/HIROX).
  There are 5 levels of evaluation, and judgment is made using the following criteria.
  -2 (Poor), -1 (Slightly Poor), 0 (Normal), 1 (Somewhat Good), 2 (Good) Time Frame: Week 0, 2, 4, 8 and week 4 after the end of intake

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Nakajima, MD, Study Chair — Ueno Asagao Clinic
Locations (1):
- Ueno Asagao Clinic, Taito-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.